CLINICAL TRIAL: NCT05925114
Title: A Phase 2, Multicenter, Randomized, Double-blind, Dose-ranging, Placebo-controlled Study to Assess the Safety and Efficacy of S-309309 in Obese Adults
Brief Title: Safety and Efficacy Study of S-309309 in Obese Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2201N1121
Record Dates: First submitted 2023-06-21; First posted 2023-06-29 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Obesity
Keywords: Body Weight; Waist; Body Mass Index (BMI)
MeSH Terms: conditions — Obesity; Body Weight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Level 1: S-309309 (Experimental): Participants will receive S-309309 (low dose) once daily for 24 weeks
  Interventions: Drug: S-309309
- Dose Level 2: S-309309 (Experimental): Participants will receive S-309309 (middle dose) once daily for 24 weeks
  Interventions: Drug: S-309309
- Dose Level 3: S-309309 (Experimental): Participants will receive S-309309 (high dose) once daily for 24 weeks
  Interventions: Drug: S-309309
- Placebo (Placebo Comparator): Participants will receive placebo once daily for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: S-309309 — Administered as oral capsules
  Arms: Dose Level 1: S-309309; Dose Level 2: S-309309; Dose Level 3: S-309309
Drug: Placebo — Administered as an oral capsule that looks identical to S-309309 capsule
  Arms: Placebo

SUMMARY:
The primary objective of this study is to understand the efficacy of S-309309 on the body weight of obese adults.

ELIGIBILITY:
Key Inclusion Criteria:

1. BMI of ≥ 30 kg/m^2 (obese) with or without comorbidities. An online BMI calculator is available at Calculate Your BMI - Standard BMI Calculator (nih.gov)
2. Stable body weight (defined as ≤ 5 kg of self-reported change) within 90 days prior to study start
3. Lifetime history of at least 1 unsuccessful dietary effort to lose body weight
4. Is a participant of non-childbearing potential (PONCBP) OR Is a participant of childbearing potential (POCBP) and using a contraceptive method that is highly effective as specified in the protocol. A POCBP must have a negative highly sensitive pregnancy test (urine or serum) before a first dose of study intervention as per protocol.

Key Exclusion Criteria:

1. Obesity of known endocrine origin (eg, untreated hypothyroidism, Cushing's syndrome)
2. Medical history or characteristics suggestive of genetic obesity
3. Any lifetime history of a suicide attempt or history of any suicidal ideation within the past year before entry into the study
4. History of documented human immunodeficiency virus (HIV) infection
5. History of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data
6. History of inflammatory conditions and autoimmune diseases
7. Males: a QT interval corrected using Fridericia's formula (QTcF) interval of > 450 msec at the Screening Visit; females: a QTcF interval > 470 msec at the Screening Visit
8. Active malignancy or history of malignancy (other than nonmelanoma skin cancer or any grade intraepithelial cervical neoplasia that has been surgically treated) within 5 years of enrollment in this study
9. A severe psychiatric condition, such as schizophrenia, bipolar disorder, or major depression in the previous 2 years before the Screening Visit, or history of treatment with antipsychotics, antidepressants, or mood stabilizers in the previous 2 years before the Screening Visit.
10. Suicidal ideation corresponding to type 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) within the past 30 days prior to the Screening Visit
11. A Patient Health Questionnaire-9 (PHQ-9) score of ≥ 15 at the Screening Visit
12. History of an eating disorder (eg, bulimia or anorexia nervosa)
13. History of drug or alcohol abuse within 5 years of the Screening Visit
14. A self-reported change in body weight > 5 kg (11 pounds [lbs]) within 90 days prior to the Screening Visit
15. Known history of treated or untreated diabetes
16. Baseline hemoglobin A1c (HbA1c) ≥ 6.5% at the Screening Visit
17. Alanine aminotransaminase (ALT) > 3 × upper limit of normal (ULN) at the Screening Visit
18. Aspartate aminotransaminase (AST) > 3 × ULN at the Screening Visit
19. Estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m^2 according to the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) at the Screening Visit
20. Chronic history of or current liver disease or known hepatic or biliary abnormalities (with the exception of nonalcoholic fatty liver disease, nonalcoholic steatohepatitis, Gilbert's syndrome or gallstones)
21. Any underlying lens opacity that affects the BCVA, or any posterior subcapsular opacity ≥ P1 based on the LOCS III, even if not impacting the BCVA
22. Marijuana use within 90 days prior to the Screening Visit
23. Use of medications that the investigator considers to be associated with weight changes within 90 days prior to the Screening Visit
24. Concomitant or previous steroid treatments (including eye-drops, inhalers, and nebulizers) for a total of ≥ 15 days during the 24 weeks prior to the Screening Visit; dermatological preparations of steroids will be allowed
25. History of or planned bariatric surgery or intra-abdominal balloon during study participation
26. Concomitant use of any dietary or herbal supplement that is indicated for weight management or maintenance of healthy weight
27. Use of drugs or substances known to be inducers or inhibitors of P-glycoprotein (P-gp) within 28 days prior to dosing
28. Received any investigational drug within 3 months of the Screening Visit
29. History of coronavirus disease 2019 (COVID-19) infection within 14 days prior to the Screening Visit or close contact with a COVID-19 patient in the 14 days prior to the Screening Visit as reported by the participant and the participant's medical history
30. Presence of HIV antibody at the Screening Visit or within 90 days prior to the Screening Visit
31. Regularly consumes excessive amounts of alcohol, defined as > 3 glasses of alcoholic beverages per day
32. Sensitivity to any of the study interventions, or components thereof, or drug or other allergy, that, in the opinion of the investigator or medical monitor, contraindicates participation in the study
33. Female study participants who have a positive urine pregnancy test at the Screening Visit
34. Female study participants who are breastfeeding
35. Poor venous access based on the investigator's judgement
36. Unable to swallow capsules
37. Hemoglobinopathy, hemolytic anemia, or chronic anemia (hemoglobin concentration < 11.5 g/dL for males, < 10.5 g/dL for females) at the Screening Visit or any other condition known to interfere with interpretation of HbA1c measurement

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2023-06-21 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-05-17 (Actual)

PRIMARY OUTCOMES:
Percent Change From Baseline in Body Weight | Baseline, Week 24

SECONDARY OUTCOMES:
Percentage of Participants Achieving a Weight Loss of ≥ 5% | Baseline to Week 24
Percentage of Participants Achieving a Weight Loss of ≥ 10% | Baseline to Week 24
Percentage of Participants Achieving a Weight Loss of ≥ 15% | Baseline to Week 24
Percentage of Participants Achieving a Weight Loss of ≥ 20% | Baseline to Week 24
Change From Baseline in Waist Circumference | Baseline, Week 24
Change From Baseline in Hip/Waist Ratio | Baseline, Week 24
Change From Baseline in BMI | Baseline, Week 24
Change From Baseline in Glucose Metabolism Parameters as Assessed by Hemoglobin A1c or Glycosylated Hemoglobin (HbA1c) | Baseline, Week 24
Change From Baseline in Glucose Metabolism Parameters as Assessed by Fasting Plasma Glucose (FPG) | Baseline, Week 24
Change From Baseline in Cardiovascular Risk Factors | Baseline, Week 24
Change From Baseline in Body Composition: Total Fat Mass as Assessed by DEXA scan | Baseline, Week 24
Change From Baseline in Body Composition: Lean Mass as Assessed by DEXA scan | Baseline, Week 24
Change From Baseline in Body Composition: Visceral Fat Mass as Assessed by DEXA scan | Baseline, Week 24
Plasma Concentration of S-309309 | Up to 24 weeks
Change From Baseline in Adiponectin | Baseline, Week 24
Change From Baseline in High Sensitivity C-reactive Protein (hsCRP) | Baseline, Week 24
Change From Baseline in Leptin | Baseline, Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Shionogi
Locations (48):
- United States (48):
  - Flourish Research - Birmingham - PPDS, Birmingham, Alabama
  - Synexus Clinical Research, Birmingham, Alabama
  - Foothills Research Center - CCT - PPDS, Phoenix, Arizona
  - National Research Institute - ClinEdge - PPDS, Los Angeles, California
  - Catalina Research Institute, Montclair, California
  - Northern California Research Corp, Sacramento, California
  - Encompass Clinical Research - ClinEdge - PPDS, Spring Valley, California
  - Chase Medical Research LLC, Waterbury, Connecticut
  - A G A Clininical Trials- HyperCore PPDS, Hialeah, Florida
  - Westside Center for Clinical Research - ERN - PPDS, Jacksonville, Florida
  - 3Sync, LLC, Lake Worth, Florida
  - Suncoast Research Group LLC - Flourish - PPDS, Miami, Florida
  - Angels Clinical Research Institute-Miami, Miami Lakes, Florida
  - Oviedo Medical Research - ClinEdge PPDs, Oviedo, Florida
  - Precision Clinical Research, Sunrise, Florida
  - Endocrine Consultants Research - Columbus - Centricity Research - HyperCore - PPDS, Columbus, Georgia
  - Javara, Inc./Privia Medical Group Georgia, LLC - Fayetteville - Javara - PPDS, Fayetteville, Georgia
  - Lifeline Primary Care - CCT-PPDS, Lilburn, Georgia
  - Flourish Research - Ravenswood - PPDS, Chicago, Illinois
  - L MARC Research Center, Louisville, Kentucky
  - Annapolis Internal Medicine, LLC, Annapolis, Maryland
  - Privia Medical Group Mid-Atlantic - Javara - PPDS, Silver Spring, Maryland
  - Boston Clinical Trials Inc. - Alcanza - HyperCore - PPDS, Boston, Massachusetts
  - ActivMed Practices & Research, Inc. - Portsmouth - Alcanza - HyperCore - PPDS, Methuen, Massachusetts
  - Be Well Clinical Studies LLC, Lincoln, Nebraska
  - Palm Research Center, Inc, Las Vegas, Nevada
  - Tryon Medical Practice - Ballantyne - Javara - PPDS, Charlotte, North Carolina
  - Lucas Research - Hickory - HyperCore - PPDS, Hickory, North Carolina
  - AES - DRS - Synexus Clinical Research US, Inc., Akron, Ohio
  - Velocity Clinical Research (Cincinnati - Ohio) - PPDS, Cincinnati, Ohio
  - Lynn Institute of East Oklahoma - ERN PPDS, Oklahoma City, Oklahoma
  - Hatboro Medical Associates PC, Hatboro, Pennsylvania
  - Medical Care, LLC, Elizabethton, Tennessee
  - Dallas Diabetes Research Center, Dallas, Texas
  - Helios CR Ins Houston - PPDS, Houston, Texas
  - Juno Research LLC, Houston, Texas
  - Edrocrine and Psychiatry Center, Houston, Texas
  - Helios CR, Inc. - Keller - PPDS, Keller, Texas
  - Vytalus Medical Group, Kingwood, Texas
  - Flourish Research, San Antonio, Texas
  - Diabetes and Gandular Disease Clinic, PA, San Antonio, Texas
  - Consano Clinical Research, San Antonio, Texas
  - AES - DRS - Synexus Clinical Research US, Inc, Murray, Utah
  - Ogden Clinic - Grand View, Roy, Utah
  - Olympus Family Medicine - CCT - PPDS, Salt Lake City, Utah
  - South Ogden Family Medicine, South Ogden, Utah
  - Charlottesville Medical Research Center, Charlottesville, Virginia
  - Manasas Clinical Research Center, Manassas, Virginia

IPD SHARING:
Plan to Share IPD: No